CLINICAL TRIAL: NCT04064723
Title: Link LCU + Lima Delta TT vs DePuy Corail + Pinnacle. A Comparative Study of Stem and Cup Fixation and Polyethylene Wear
Brief Title: A Comparative Study of Stem and Cup Fixation and Polyethylene Wear
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCU-DeltaTT
Record Dates: First submitted 2019-04-23; First posted 2019-08-22 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Osteoarthritis; Total hip arthroplasty; Uncemented total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Control: Corail femoral stem and Pinnacle cup with Marathon XLPE neutral liner (DePuy Orthopaedics).
  Study: LCU femoral stem (Waldemar Link GmbH) and Delta TT cup with Neutral XLPE liner (Lima Corporate).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem components (Active Comparator): Randomization between two stem components. LCU or Corail stem.
  Interventions: Device: Randomization between prosthetic components
- Cup components (Active Comparator): Randomization between two cup components. DeltaTT or Pinnacle cup.
  Interventions: Device: Randomization between prosthetic components

INTERVENTIONS:
Device: Randomization between prosthetic components — Patients are randomized between two types of stem components and two types of cup components in total hip arthroplasty. Thus randomized between 4 different groups.

SUMMARY:
A randomized controlled study comparing two types of cementless femoral stems (LCU and Corail) and two types of acetabular components (DeltaTT and Pinnacle Duofix) in primary total hip arthroplasty. Primary outcome are component migration measured by RSA, wear and patient reported outcome. Patients are evaluated up to 15 years postoperatively.

DETAILED DESCRIPTION:
Material Patients The study will be conducted according to GCP, (Good Clinical Practice). Potential clinical study participants will be identified from the THR waiting list of Umeå University Hospital. The enrolment process will involve a review of the patient history from the medical records in order to match available patient details with the inclusion/exclusion criteria (see below). Patients considered suitable for potential study enrolment will be contacted by a member of the research team to ascertain their level of interest in participating in this study.

Once verbal and written informed consent is provided a medical profile will be taken.

Inclusion criteria:

Primary or secondary osteoarthritis of the hip Male and non-pregnant female patients aged 18 to 70 years of age Type A or B femur Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up

Exclusion criteria BMI under 18 and over 35 Inflammatory arthritis Osteoporosis Paget's disease Grossly abnormal hip anatomy (severe dysplasia) Previous operations in the same hip Presence of malignancy Patients who, as judged by the surgeon, are mentally incompetent or are reasonable unlikely to be compliant with the requirements of the study Patient is female of child-bearing age and not taking contraceptive precautions

Implants Control: Corail femoral stem and Pinnacle cup with Marathon XLPE neutral liner (DePuy Orthopaedics), Bilolox delta ceramic femoral head 32 mm Study: LCU femoral stem (Waldemar Link GmbH) and Delta TT cup with Neutral XLPE liner (Lima Corporate), Biolox delta ceramic femoral head 32 mm.

For both designs a 28 mm femoral head will be used when cup size (< 48 mm) precludes the use of larger head.

The stems will be fitted with 2 tantalum markers by the surgeon at the operation. One tantalum marker will be fixed in a small PEEK tower that will be screwed in at the shoulder of the stem. Another tantalum marker will be cemented at the tip of the stem before insertion. The PE liners will be fitted with tantalum beads by the surgeon at the time of surgery.

The shell of the Delta TT cup will have 2 to 3 tantalum markers attached to its outer surface. This process will be done by a subcontractor to the manufacturer.

Randomization Stratification for gender will be done. Within each stratum there will be block randomization with 8 permutations in each block, each permutation will be either LCU+Delta TT, LCU+Pinnacle, Corail+Delta TT, or Corail+Pinnacle. The randomization plan generator available at www.randomization.com will be used to create the randomization which will then be put in consecutively numbered sealed envelopes, one series for each stratum. The envelopes will be located in a locked cabinet at the research nurse office. Due to logistic reasons it will not be possible to open the sealed envelope at the time for surgery. Instead the surgeon the day before surgery calls the research nurse who opens the envelope and assigns the patient name to that randomization. This procedure will ensure that correct instrumentation and implants will be available for surgery.

Operative technique All patients will be operated through a postero-lateral approach. The height of the resection of the collum femoris is determined by preoperative templating. The acetabulum is prepared by reaming in 2 mm increments until a good bone contact is established. The press fit is tested with a trial cup. The recommendation is to use a cup the same size as the last reamer, line-to-line. The aim is 35 to 45 degrees of abduction and 15-20 degrees of anteversion. Additional screws are only used if surgeon considers that absolutely necessery. As standard a neutral liner is used routinely. If no sufficient stability of the hip is established with the neutral liner, a 20° lipped liner is used as a compromise solution. In case of acetabular fracture additional screws may be used but the patient is then excluded from the study.

The femoral canal is opened with a box chisel and a straight rasp is used for identifying the center of the femoral canal. Preparation is always started with the smallest broach. The size of the broach is increased until rotational stability in the preoperatively planed height is reached. A trial reduction, including testing of hip stability, is then performed. When adequate leg length, offset and stability is reached the definitive stem is inserted. If a femoral fracture occurs during operation a collared stem is used together with cerclage wiring and the patient will be excluded from the study. The ceramic head is assembled on to the properly cleaned taper with one firm blow.

9 Tantalum markers will be inserted into the bone of the pelvis around acetabulum and 9 in the proximal femur using a special inserter. Tantalum markers will also be inserted into the polyethylene liner and, in case of Delta TT cup, into the outer surface of the metal cup. Finally 1 tantalum marker affixed to a purposely made PEEK tower will screwed onto the shoulder of the femoral stem and 1 marker cemented onto the tip of the stem.

Intra op measurements Clinical quality of cup and stem insertion (surgeon's judgement): excellent, good, doubtful Degrees of femoral internal rotation at 90 degrees of hip flexion at time for subluxation of femoral head.

Size of last cup and stem reamer/broach All implant parameters

RSA Measurement of polyethylene wear, stem and cup migration and liner-shell fixation is measured with RSA within one week postop, and thereafter at 1½ mo, 3 mo, 12 mo, 24 mo, 5y, 10 y, and 15 y postoperatively.

RSA has been used for implant research for over 30 years, with several hundreds of publications, and is considered the golden standard for this type of research.

At the time of operation tantalum spheres/markers (diameter 1 mm) are inserted into proximal femur, periacetabular area and in the polyethylene liner in a standardized manner. The femoral components will be equipped with 2 tantalum spheres in prefabricated cases.

Conventional x rays AP pelvis and AP + lateral of affected hip will be obtained preop. (for templating), within one week postop. (check and measurement of alignment) and at 12 mo, 24 mo, 5 y, 10 y and 15 y (for determination of osseointegration and osteolysis/stress shielding).

Computed tomography (CT) CT of the pelvis around the cup will be performed 24 months and 5 or 10 years postoperatively to determine potential acetabular osteolysis / bone resorption.

Clinical evaluation Patient reported outcome measures: HOOS, Harris Hip Score, EQ5D, EQ5D VAS, SF-36 and UCLA activity score will be obtained preoperatively, and at all postoperative follow-ups.

Serological measurements Level of serum titanium will be measured preoperative, and at 12 mo, 24 mo, 5y, 10 y, and 15 y postoperative

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary osteoarthritis of the hip
* Male and non-pregnant female patients aged 18 to 70 years of age
* Type A or B femur
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up

Exclusion Criteria:

* BMI under 18 and over 35
* Inflammatory arthritis
* Osteoporosis
* Paget's disease
* Grossly abnormal hip anatomy (severe dysplasia)
* Previous operations in the same hip
* Presence of malignancy
* Patients who, as judged by the surgeon, are mentally incompetent or are reasonable unlikely to be compliant with the requirements of the study
* Patient is female of child-bearing age and not taking contraceptive precautions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Cup Migration | 1-15 years
  Migration measured in millimetres per year with radiostereometric (RSA) analysis of radiographs. Radiostereometric analysis (RSA) is a stereo X-ray technique used in clinical research studies to evaluate micro-motion and wear of orthopaedic implants within bone. The method has a high accuracy and precision. Technical requirements include the need for implanted marker beads and radiograph view angles determined by a calibration cage.
Femoral stem migration | 1-15 years
  Migration measured in millimetres per year with radiostereometric (RSA) analysis of radiographs.
Wear | 1-15 years
  The size of the femoral component penetration into the polyethylene measured in millimeters per year and the volumetric annual wear millimetres with radiostereometric (RSA) analysis of radiographs.

SECONDARY OUTCOMES:
Movement between liner and acetabular components | 1-15 years
  Movements between the polyethylene liner and the metal shell of the Delta TT millimetres with radiostereometric (RSA) analysis of radiographs measured in millimeters per year.
Patient reported outcome measurement | 1-15 years
  Hip disability and Osteoarthritis Outcome Score is a disease specific patient reported outcome measures ranging from 0-100 points. Obtained preoperatively, and at all postoperative follow-ups 6 weeks, 3, 12 months, 2, 5, 10 and 15 years.
Harris Hip Score | 1-15 years
  Harris Hip score is a patient reported outcome measure which include questions regarding the function of the treated hip. Obtained preoperatively, and at all postoperative follow-ups 6 weeks, 3, 12 months, 2, 5, 10 and 15 years.
EQ5D | 1-15 years
  A general health related quality of life questionnaire of which a score i calculated (-0,594-1.0). Obtained preoperatively, and at all postoperative follow-ups 6 weeks, 3, 12 months, 2, 5, 10 and 15 years.
Visual Analog Scale | 1-15 years
  Visual Analog Scale (0-100 points) obtained preoperatively, and at all postoperative follow-ups 6 weeks, 3, 12 months, 2, 5, 10 and 15 years.
University of California, Los Angeles (UCLA) activity scale | 1-15 years
  Patient reported outcome measure for evaluating activity University of California, Los Angeles (UCLA) activity scale (0-10). Obtained preoperatively, and at all postoperative follow-ups 6 weeks, 3, 12 months, 2, 5, 10 and 15 years.
Short Form Health Survey | 1-15 years
  Short Form Health Survey (0-100 points) is a general health related quality of life patient reported outcome measure Obtained preoperatively, and at all postoperative follow-ups 6 weeks, 3, 12 months, 2, 5, 10 and 15 years.

CONTACTS AND LOCATIONS:
Overall Officials: Volker TC Otten, M.D., Ph.D, Principal Investigator — Umeå University
Locations (1):
- Volker TC Otten, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joglekar SB, Rose PS, Lewallen DG, Sim FH. Tantalum acetabular cups provide secure fixation in THA after pelvic irradiation at minimum 5-year followup. Clin Orthop Relat Res. 2012 Nov;470(11):3041-7. doi: 10.1007/s11999-012-2382-8. PMID 22576931
- [Background] Goriainov V, Jones A, Briscoe A, New A, Dunlop D. Do the cup surface properties influence the initial stability? J Arthroplasty. 2014 Apr;29(4):757-62. doi: 10.1016/j.arth.2013.07.007. Epub 2013 Nov 22. PMID 24269067
- [Background] Engh CA Jr, Stepniewski AS, Ginn SD, Beykirch SE, Sychterz-Terefenko CJ, Hopper RH Jr, Engh CA. A randomized prospective evaluation of outcomes after total hip arthroplasty using cross-linked marathon and non-cross-linked Enduron polyethylene liners. J Arthroplasty. 2006 Sep;21(6 Suppl 2):17-25. doi: 10.1016/j.arth.2006.05.002. PMID 16950057
- [Background] Campbell D, Mercer G, Nilsson KG, Wells V, Field JR, Callary SA. Early migration characteristics of a hydroxyapatite-coated femoral stem: an RSA study. Int Orthop. 2011 Apr;35(4):483-8. doi: 10.1007/s00264-009-0913-z. Epub 2009 Dec 13. PMID 20012862
- [Background] Karrholm J, Herberts P, Hultmark P, Malchau H, Nivbrant B, Thanner J. Radiostereometry of hip prostheses. Review of methodology and clinical results. Clin Orthop Relat Res. 1997 Nov;(344):94-110. PMID 9372762
- [Background] Baad-Hansen T, Kold S, Nielsen PT, Laursen MB, Christensen PH, Soballe K. Comparison of trabecular metal cups and titanium fiber-mesh cups in primary hip arthroplasty: a randomized RSA and bone mineral densitometry study of 50 hips. Acta Orthop. 2011 Apr;82(2):155-60. doi: 10.3109/17453674.2011.572251. Epub 2011 Mar 25. PMID 21434845
- [Background] Bitsch RG, Loidolt T, Heisel C, Ball S, Schmalzried TP. Reduction of osteolysis with use of Marathon cross-linked polyethylene. A concise follow-up, at a minimum of five years, of a previous report. J Bone Joint Surg Am. 2008 Jul;90(7):1487-91. doi: 10.2106/JBJS.F.00991. PMID 18594097
- [Background] Madanat R, Makinen TJ, Aro HT, Bragdon C, Malchau H. Adherence of hip and knee arthroplasty studies to RSA standardization guidelines. A systematic review. Acta Orthop. 2014 Sep;85(5):447-55. doi: 10.3109/17453674.2014.934187. Epub 2014 Jun 23. PMID 24954489
- [Background] van der Voort P, Pijls BG, Nieuwenhuijse MJ, Jasper J, Fiocco M, Plevier JW, Middeldorp S, Valstar ER, Nelissen RG. Early subsidence of shape-closed hip arthroplasty stems is associated with late revision. A systematic review and meta-analysis of 24 RSA studies and 56 survival studies. Acta Orthop. 2015;86(5):575-85. doi: 10.3109/17453674.2015.1043832. PMID 25909455
- [Background] Wolf O, Mattsson P, Milbrink J, Larsson S, Mallmin H. Periprosthetic bone mineral density and fixation of the uncemented CLS stem related to different weight bearing regimes: A randomized study using DXA and RSA in 38 patients followed for 5 years. Acta Orthop. 2010 Jun;81(3):286-91. doi: 10.3109/17453674.2010.487238. PMID 20446828
- [Background] Drobniewski M, Borowski A, Synder M, Sibinski M. Results of total cementless hip joint arthroplasty with Corail stem. Ortop Traumatol Rehabil. 2013 Jan-Feb;15(1):61-8. doi: 10.5604/15093492.1032797. PMID 23510822
- [Background] Louboutin L, Viste A, Desmarchelier R, Fessy MH. Long-term survivorship of the Corail standard stem. Orthop Traumatol Surg Res. 2017 Nov;103(7):987-992. doi: 10.1016/j.otsr.2017.06.010. Epub 2017 Aug 1. PMID 28778624
- [Background] Buttaro MA, Onativia JI, Slullitel PA, Andreoli M, Comba F, Zanotti G, Piccaluga F. Metaphyseal debonding of the Corail collarless cementless stem: report of 18 cases and case-control study. Bone Joint J. 2017 Nov;99-B(11):1435-1441. doi: 10.1302/0301-620X.99B11.BJJ-2017-0431.R1. PMID 29092981